CLINICAL TRIAL: NCT02575872
Title: The Effectiveness of a Comprehensive Physical Activity Behavioral Intervention on Underserved Diverse Obese Endometrial Cancer Survivors
Brief Title: Physical Activity Behavioral Intervention in Obese Endometrial Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nicole Nevadunsky, Principal Investigator, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2013-2167; NCI-2014-01510 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-2167 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Stage IA Uterine Corpus Cancer; Stage IB Uterine Corpus Cancer; Stage II Uterine Corpus Cancer; Stage IIIA Uterine Corpus Cancer; Stage IIIB Uterine Corpus Cancer; Stage IIIC Uterine Corpus Cancer; Stage IVA Uterine Corpus Cancer; Stage IVB Uterine Corpus Cancer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Intervention (Experimental): Participants partake in 30 minutes of group discussions regarding physical activity behavior followed by 60 minutes of moderate-intensity exercise comprised of 5 minutes warm-up, 25 minutes cardiovascular training, 20 minutes of resistance training exercises using body weight and exercise band, and 10 minutes of cool-down and stretching once weekly for 12 weeks. Participants also complete a brisk walk for 90 minutes per week outside of class for 12 weeks.
  Interventions: Behavioral: Exercise Intervention
- wait-list for intervention (No Intervention): Participants receive a handout indicating the importance of physical activity and improved nutrition for health outcomes. After 12 weeks, patients are invited to participate in the physical behavior intervention as in Group I.

INTERVENTIONS:
Behavioral: Exercise Intervention — Participate in physical activity behavioral intervention
  Arms: Exercise Intervention

SUMMARY:
This randomized clinical trial studies a physical activity behavioral intervention in obese endometrial cancer survivors. Learning about physical activity behavior while participating in a fitness class may help increase physical activity and improve the quality of life of obese endometrial cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of a 12-week behavior/exercise intervention on moderate-vigorous physical activity (> 150 minutes) among ethnically diverse endometrial cancer survivors.

SECONDARY OBJECTIVES:

I. To determine the effects of a 12-week behavior/exercise intervention on body composition among ethnically diverse endometrial cancer survivors.

TERTIARY OBJECTIVES:

I. To determine the effects of a 12-week behavior/exercise intervention for ethnically diverse endometrial cancer survivors on physical function and quality-of-life.

II. To determine the most important behavioral variables for predicting physical activity adherence.

III. To determine the most significant facilitators and barriers to adherence during the 12-week intervention.

IV. To compare the thematic differences between high-adherence and low-adherence participants and qualitatively assess the strengths and weaknesses of the 12-week intervention.

OUTLINE: Participants are randomized to 1 of 2 groups

GROUP I: Participants partake in 30 minutes of group discussions regarding physical activity behavior followed by 60 minutes of moderate-intensity exercise comprised of 5 minutes warm-up, 25 minutes cardiovascular training, 20 minutes of resistance training exercises using body weight and exercise band, and 10 minutes of cool-down and stretching once weekly for 12 weeks. Participants also complete a brisk walk for 90 minutes per week outside of class for 12 weeks.

GROUP II: Participants receive a handout indicating the importance of physical activity and improved nutrition for health outcomes. After 12 weeks, patients are invited to participate in the physical behavior intervention as in Group I.

After completion of study, participants are followed up at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent form signed and dated by the subject
* English and/or Spanish speaking
* History of endometrial cancer stage I-IV > 6 months < 5 years, not currently receiving cancer treatment
* Overweight (body mass index [BMI] >= 30)
* Eastern Cooperative Oncology Group performance status (PS) of 0 - 2
* Medically capable of performing moderate intensity exercise

Exclusion Criteria:

* Must not have engaged in a regular (> 3x/week, physical activity program in the last 6 months)
* Medical contraindication to exercise

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Proportion of participants completing at least 150 minutes of moderate-vigorous physical activity, assessed by the Yale Physical Activity Survey (YPAS) | 12 weeks
  Data will be analyzed using Pearson Chi-square test.

SECONDARY OUTCOMES:
Barrier avoidance/coping, measured using 5 point Likert scales | Up to 12 weeks
  Multiple logistic regression analysis will be used to examine the association of the Social Cognitive Theory behavior variables to physical activity, adjusting for potential confounders.
BMI | Up to 12 weeks
  Will be analyzed using student t-test. When the data are non-normal, investigators will use appropriate nonparametric tests.
Change in ability to perform activities of daily living, assessed with the YPAS | Baseline to 12 weeks
  Will be analyzed using student t-test. When the data are non-normal, investigators will use appropriate nonparametric tests.
Change in sedentary time, assessed with the YPAS | Baseline to 12 weeks
  Will be analyzed using student t-test. When the data are non-normal, investigators will use appropriate nonparametric tests.
Exercise efficacy, measured using 5 point Likert scales | Up to 12 weeks
  Multiple logistic regression analysis will be used to examine the association of the Social Cognitive Theory behavior variables to physical activity, adjusting for potential confounders.
Fatigue, assessed by the FACT-Fatigue | Up to 12 weeks
  Will be analyzed using student t-test. When the data are non-normal, investigators will use appropriate nonparametric tests.
Outcome expectations, measured using 5 point Likert scales | Up to 12 weeks
  Multiple logistic regression analysis will be used to examine the association of the Social Cognitive Theory behavior variables to physical activity, adjusting for potential confounders.
Physical function score | Up to 12 weeks
  Will be analyzed using student t-test. When the data are non-normal, investigators will use appropriate nonparametric tests.
Quality of life, assessed by the Functional Assessment of Cancer Therapy (FACT)-Endometrial Cancer | Up to 12 weeks
  Will be analyzed using student t-test. When the data are non-normal, investigators will use appropriate nonparametric tests.
Self-regulation, measured using 5 point Likert scales | Up to 12 weeks
  Multiple logistic regression analysis will be used to examine the association of the Social Cognitive Theory behavior variables to physical activity, adjusting for potential confounders.
Social support, measured using 5 point Likert scales | Up to 12 weeks
  Multiple logistic regression analysis will be used to examine the association of the Social Cognitive Theory behavior variables to physical activity, adjusting for potential confounders.
Waist circumference | Up to 12 weeks
  Will be analyzed using student t-test. When the data are non-normal, investigators will use appropriate nonparametric tests.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Nevadunsky, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Derived] Agnew H, Kitson S, Crosbie EJ. Interventions for weight reduction in obesity to improve survival in women with endometrial cancer. Cochrane Database Syst Rev. 2023 Mar 27;3(3):CD012513. doi: 10.1002/14651858.CD012513.pub3. PMID 36971688